CLINICAL TRIAL: NCT04394949
Title: Securing Employment and Economic Keys to Stability (SEEKS)
Brief Title: Securing Employment and Economic Keys to Stability for Persons With Disabilities
Acronym: SEEKS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Communication Institute International, Inc. (Industry)
Collaborators: Colorado School of Public Health (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Yvonne Kellar-Guenther, Senior Research Associate, Communication Institute International, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DPCP19000085
Record Dates: First submitted 2020-04-13; First posted 2020-05-20 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Employment
Keywords: employment; education; persons with disabilities; social connection
MeSH Terms: interventions — Multicenter Studies as Topic

STUDY DESIGN:
Intervention Model Description: Randomize at the participant level (individual level block) for larger centers that have multiple Independent Living (IL) Specialists. Participant will be randomly assigned to work with a staff who is trained in the experimental services or usual care. CILs that cannot accommodate both the experimental services and usual care, cluster randomization will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Business as Usual Arm (Active Comparator): Consumers will usual care
  Interventions: Other: Usual Care
- Experimental Arm (Experimental): Center for Independent Living (CIL) consumers randomized to work with a group of CIL employees who received training in SOAR, Customized Employment, Supported Employments, and Benefits Planning (CWIC).
  Interventions: Behavioral: Center for Independent Living SEEKS Team

INTERVENTIONS:
Behavioral: Center for Independent Living SEEKS Team — Center for Independent Living (CIL) consumers randomized to work with a group of CIL employees who received training in SOAR, Customized Employment, Supported Employments, and Benefits Planning (CWIC).
  Arms: Experimental Arm
Other: Usual Care — Consumers will get same CIL services they would get if they were not enrolled in the study.
  Arms: Business as Usual Arm

SUMMARY:
There is a myth that if a person is applying for SSI/SSDI he cannot seek employment. This goal of this research is to learn if a new model of service can lead to employment, increase in gross wages, and a decrease in social isolation for persons with disabilities who work with Centers for Independent Living on applying for SSI/SSDI benefits. The researchers want to compare the services these centers typically offer these consumers to a new model - a team trained in (1) the SOAR model for SSI/SSDI application assistance, (2) certified benefits planning training, (3) customized employment training, and (4) individual employment placement services.

DETAILED DESCRIPTION:
Hypotheses and Specific Aims: The goal of the SEEKS research project is to increase employment for adult persons (ages 18-60 years of age) with disabilities who get services from a Center for Independent Living (CIL), increase gross income, and/or reduce social isolation. Our broad grant objectives are:

Objective 1: Connect persons with disabilities applying for Supplemental security Income (SSI)/Social Security Disability Insurance (SSDI) with competitive employment.

Objective 1a: Train CIL staff to utilize SSI/SSDI Outreach, Access, and Recovery (SOAR) strategies.

Objective 1b: Train CIL staff in Customized Employment

Objective 2: Provide benefits counseling to persons with disabilities applying for SSI/SSDI.

Objective 2a: Provide Community Work Incentives Coordinators (CWIC) Training to CIL staff so they can provide benefit counseling to persons with disabilities applying for SSI/SSDI.

Objective 3: Increase connections for persons with disabilities who are seeking independent living services.

To meet these objectives, the investigators are conducting a randomized control trial where CIL consumers who agree to be in the study will be randomized to work with a group of CIL employees who received training in SOAR, Customized Employment, Supported Employments, and Benefits Planning (CWIC) (Treatment Group) to consumers working with CIL employees who will offer business as usual (Control Group). The hypotheses are:

H1: Significantly more participants in the Experimental Services Group will be employed (competitive employment) than participants in the Usual Care Group at the end of the project.

H1a: Significantly more participants in the Experimental Services Group will be in employment greater than substantial gainful activity (SGA) at the end of the program than participants in the Usual Care Group.

H2: Participants in the Experimental Services Group will report a significantly higher gross income (wages and/or benefits) at the end of the program than participants in the Usual Care Group.

H2a - Significantly more participants in the Experimental Services Group will report a higher level of satisfaction with their income at the end of the program than participants in the Usual Care Group.

H3: Participants in the Experimental Services Group will report a significantly greater change in social connection scores from when they entered the program to the end of the program than participants in the Usual Care Group.

H3a: Participants in the Experimental Services Group will significantly show a greater change in highest education obtained from when they entered the program to the end of the program than participants in the Usual Care Group.

Background and Significance:

Overview of Intervention Being Tested. This project is comparing two service delivery models to determine which results in increased competitive integrative employment, increase gross income, and increased social inclusion for persons with disabilities aged 18-60 years who are interested in applying for Supplemental Security Income (SSI)/Social Security Disability Insurance (SSDI) benefits. Both groups will include consumers who work with one of the participating Centers for Independent Living (CILs) in Colorado. CIL staff working with the intervention group will be trained in using the following:

* SOAR strategies,
* the Individual Placement and Support (IPS) model and
* competitive employment (CE) strategies and
* comprehensive benefits counseling (CWIC). CIL staff working with the control group will deliver their usual CIL services.

While SOAR strategies, Employment Services using the IPS model and CE strategies, and comprehensive benefits counseling have all been shown to be impactful on employment individually, there has not been a test of an intervention that uses and integrates all three strategies for adults with disabilities who are working with CILs and range in age from 18 to 60 years of age.

CILs work to support community living and independence for persons with disabilities. CILs believe work experience, post-secondary education, and reduced social isolation are all important. As a result, this program will look at how training CIL staff in SOAR strategies, the IPS model, CE strategies, and comprehensive benefits counseling will impact not just employment but also pursuing post-secondary education and increased connection to others.

Summary of previously published data and pilot studies on need of the target population. Nationally, data on employment rates from 2017 illustrate a large discrepancy, 40%, between the employment rates of people with disabilities compared to those without disabilities. More specifically, the employment rate for those 18-64 without disabilities is 77.2% versus the same age group of individuals with disabilities at 37%. Even though the gap is not quite as large in Colorado, 2019 data shows that the employment for those without disabilities is 66.3% compared to those with disabilities at 19.3%. This data reveals a rather large 35.1% lower employment rate for individuals with disabilities in Colorado.

In examining other documented characteristics comparing Coloradans with disabilities to those without, there are alarming differences. For example, poverty data in Colorado reveals that there are 70,811 individuals with disabilities who live in poverty. This is 22.8% of the disability population 18-64 years old. This is high compared to the same age group without disabilities, 285,268 or 9.1% of persons who do not have a disability live in poverty. Once again there is a higher rate of poverty for individuals with disabilities by 13.7%. Although the gap is not quite as wide for veterans, the poverty rate for veterans with disabilities is 6% higher than those without.

One reason the poverty level may be higher for persons with disabilities is that there are 45,852 Supplemental Security Income (SSI) recipients in Colorado ages 18-64. In 2016, the national approval rate for SSI/SSDI applications (medical decisions- all ages) was 29.8%. This means that for every 10 SSI applications submitted to SSA (Social Security Administration) only about 3 SSI applications are approved. When taking into account another 114,954 Social Security Disability Insurance (SSDI) beneficiaries identified in the 2018 Annual Disability Statistics Compendium as of December 2017, 20% of the disability population in Colorado is receiving SSA disability benefits.

Anand and Ben-Shalom conducted a study where they examined SSA administrative data to identify the most common paths followed by new SSDI and SSI recipients over a 10 year period after first award. These authors reported that 80% of SSDI first beneficiaries and 53% of SSI recipients either achieved no additional employment milestones after achieving benefits or the milestone reached was death or full retirement age. In other words, once these recipients received SSI or SSDI, movement toward employment either stopped or was considerably delayed.

Not working can be extremely problematic. Not only does it mean the SSI and SSDI recipients will live in poverty, it also increases health risks. Unemployment can lead to increased mental distress, social disconnection, increased substance use and physical illness. Some of the modifiable risks included social isolation, unemployment and poverty. These are areas that need to be addressed and can be addressed in Colorado through collaboration and realignment of Colorado systems providing services to individuals with disabilities such as the Center for Independent Living system.

Preliminary Studies/Progress Report:

The SEEKS intervention will utilize a number of documented promising practices and evidence-based practices to achieve the outcomes that the investigators are testing in our hypotheses. Over the years, the federal government has funded research and demonstration projects to test strategies to improve employment outcomes for people with disabilities. Typically, these demonstration strategies focused on either redirecting individuals from applying for Social Security Administration disability benefits as adults or assisting those already receiving SSA disability benefits to find employment. Specifically, two such notable projects are SSA's Youth Transition Demonstration and the Promoting Readiness of Minors in SSI Demonstration aimed to improve employment outcomes and decrease the benefit receipt rate for youth that are receiving or at risk of receiving SSI payments. Although both models have notable successes, there are elements of these models that do not address some of the fundamental needs of people with disabilities such as economic stability and community participation. Ergo, SEEKS targets people applying for SSA disability benefits while concurrently receiving services from an employment specialist to obtain employment and a comprehensive benefits planner. This model combines the expectation that people with disabilities can contribute to the business bottom line in the competitive, integrated workforce, but also seeks to address limited economic resources experienced by people with disabilities.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-60 years of age,
* have a disability (as defined the Centers for Independent Living federal reporting guidelines)
* be a consumer working with a Colorado Independent Living Center to apply for SSI/SSDI
* agree to work with the Division of Vocational Rehabilitation

Exclusion Criteria:

* Does not work with the Centers for Independent Living
* Does not agree to provide data every 6 months.
* Not own legal guardian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Employed in Competitive Integrative Employment | Baseline
  if employed in competitive integrated employment at time of data collection (yes/no)
Employed in Competitive Integrative Employment | Six Month Update
  if employed in competitive integrated employment at time of data collection (yes/no)
Employed in Competitive Integrative Employment | Yearly Update
  if employed in competitive integrated employment at time of data collection (yes/no)
Employed in Competitive Integrative Employment | 18 month update
  if employed in competitive integrated employment at time of data collection (yes/no)
Employed in Competitive Integrative Employment | 2 year update
  if employed in competitive integrated employment at time of data collection (yes/no)

SECONDARY OUTCOMES:
Education Level | Baseline
  education level when entering program
Change in Education Level | Six month
  has participant completed more education, including vocational rehabilitation
Change in Education Level | One year
  has participant completed more education, including vocational rehabilitation
Change in Education Level | 18 months
  has participant completed more education, including vocational rehabilitation
Change in Education Level | Two years
  has participant completed more education, including vocational rehabilitation
Gross Income Level | baseline
  Income including wages and benefits
Change in Gross Income Level | six months
  Looking for increased income including wages and benefits
Change in Gross Income Level | one year
  Looking for increased income including wages and benefits
Change in Gross Income Level | 18 months
  Looking for increased income including wages and benefits
Change in Gross Income Level | two years
  Looking for increased income including wages and benefits
Increased Personal Connections | baseline
  Interaction with others outside the home, if at desired level. Participants will indicate if they are able to build friendships, feel included in community, attend organized groups, socialize with friends, neighbors, other students, or co-workers as often as they want. The items are based off the Indicators for Social Isolation Social Participation subscale and then expanded for this study based on feedback from peer advisory committee.
Change in Increased Personal Connections | six months
  Interaction with others outside the home, if at desired level
Change in Increased Personal Connections | one year
  Interaction with others outside the home, if at desired level
Change in Increased Personal Connections | 18 months
  Interaction with others outside the home, if at desired level
Change in Increased Personal Connections | two years
  Interaction with others outside the home, if at desired level

CONTACTS AND LOCATIONS:
Locations (1):
- Yvonne Kellar-Guenther, Littleton, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be shared. Data will be at the individual level.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Anand P, Ben-Shalom Y. Pathways Taken by New Social Security Disability Insurance and Supplemental Security Income Awardees. Journal of Disability Policy Studies, 2018; 29(3), 153-165. https://doi.org/10.1177/1044207318779987
- See also: 1. Link to 2017 Disability Annual Report — https://disabilitycompendium.org/sites/default/files/user-uploads/2017_AnnualReport_2017_FINAL.pdf
- See also: 3. 2018 Annual Disability Statistics Compendium — https://disabilitycompendium.org/sites/default/files/user-uploads/2018_Compendium_Accessible_AbobeReaderFriendly.pdf
- See also: 7. Unemployment and mental health. — https://www.iwh.on.ca/summaries/issue-briefing/unemployment-and-mental-health